CLINICAL TRIAL: NCT05268250
Title: Remedy to Diabetes Distress (R2D2): A Scalable Screen to Treat Program for School-age Families
Acronym: R2D2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Susana Patton, Principal Research Scientist, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1687888
Record Dates: First submitted 2022-02-16; First posted 2022-03-07 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R2D2 mHealth treatment for diabetes distress (Experimental): This is a mHealth supported, cognitive behavioral treatment for parents and school-age children who were identified with clinically relevant levels of diabetes distress as part of a clinic screening program
  Interventions: Behavioral: R2D2 mHealth intervention
- Standard Care Control (No Intervention): Parents and school-age children who were identified with clinically relevant levels of diabetes distress as part of a clinic screening program will receive local resources (print or electronic).

INTERVENTIONS:
Behavioral: R2D2 mHealth intervention — R2D2 mHealth treatment will use cognitive behavioral therapy, mindfulness, and behavioral activation strategies
  Arms: R2D2 mHealth treatment for diabetes distress

SUMMARY:
This R01 is in response to RFA-DK-19-021, Treating Diabetes Distress to Improve Glycemic Outcomes in Type 1 Diabetes. The objective is to test the feasibility and acceptability of a novel, practical, and potentially scalable screen to treat program for diabetes distress in families of school-age children with T1D (called Remedy to Diabetes Distress [R2D2]) and to test the initial efficacy of R2D2 to reduce diabetes distress to improve children's glycemic control.

DETAILED DESCRIPTION:
Only 22% of school-age children with type 1 diabetes (T1D) achieve an HbA1c of <7.5% while the majority of school-age children who exceed this target are at higher risk for T1D-related complications. Achieving optimal T1D self-care is the only direct pathway to better HbA1c and even with the addition of modern therapeutic modalities (e.g., hybrid closed loop), it is a complex, time-consuming, and relentless task. School-age children cannot effectively manage T1D alone and require help from their parents to participate in daily T1D self-care. The research suggests that both parents and youth with T1D are vulnerable to Diabetes Distress (DD) and the American Diabetes Association (ADA) Standards of Care recommend ongoing assessment of DD in youth (starting at 7-8-years-old) and their caregiver during routine diabetes clinic visits. Unfortunately, while DD screening may be an ADA Care Standard, there are no practical treatment options for clinics to adopt to treat DD in school-age families in the case of positive screens. The researchers submit this new R01 in response to RFA-DK-19-021, Treating Diabetes Distress to Improve Glycemic Outcomes in Type 1 Diabetes. Our objective is to test the feasibility and acceptability of a novel, practical, and potentially scalable screen to treat program for DD in families of school-age children with T1D (called Remedy to Diabetes Distress [R2D2]) and to test the initial efficacy of R2D2 to reduce DD to improve children's glycemic control. To enhance scientific rigor, the researchers plan to use the ORBIT model for behavioral intervention development to guide the study design. The specific aims are: 1) Define feasibility and acceptability of our new screen to treat program (R2D2) for DD in school-age families, and 2) Establish initial efficacy of R2D2 to reduce parent and child DD to improve child glycemic control. The researchers propose to address these Aims through an iterative process and multiple projects to complete the necessary formative research to design, build, and prepare to implement R2D2. The researchers then propose to complete a Pilot randomized controlled trial of their R2D2 screen to treat program, testing for its initial efficacy based on child HbA1c and time in range (primary outcomes) and parent and child DD and resilience, and T1D self-care (secondary outcomes; Phase 2b: Pilot, n=180). The impact of the proposed R01 is high because it addresses a critical need for practical and evidence-based solutions for screening and treating DD in families of school-age children, heretofore an understudied patient subgroup. The researchers believe our study optimally responds to the FOA because the research team is multidisciplinary (anchored by a partnership between behavioral science and diabetology), and their R2D2 screen to treat program reflects a practical team approach that can realistically occur in clinic and scale to other centers.

ELIGIBILITY:
Inclusion Criteria:

* child age between 8-12 years, physician confirmed T1D diagnosis,
* either the child or the parent or both the child and parent report diabetes distress levels at or above clinical cut-points,
* child is on an intensive insulin regimen (pump or MDI).

Exclusion Criteria:

* children on a conventional insulin regimen, children and/or parents who do not report diabetes distress levels at or above the clinical cut-points,
* children who have an allergy or sensitivity to the adhesive and/or skin preparation used for CGM, children with a comorbid chronic condition (e.g., renal disease),
* children and parents who do not speak English.

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
youth glycated hemoglobin (HbA1c) | week 0, week 13
  proxy measure of average glycemic levels over 10-12 weeks
youth time in range | week 0, week 13
  based on continuous glucose levels, the percentage of time spent between 70-180mg/dl

SECONDARY OUTCOMES:
Problem Areas in Diabetes-Child (PAID-C) | week 0, week 13
  validated child report of diabetes distress; range: 11-66, higher scores reflect greater distress
Parent Problem Areas in Diabetes-Child (P-PAID-C) | week 0, week 13
  validated parent report of diabetes distress; range 16-96, higher scores reflect greater distress
Diabetes Strengths and Resilience | week 0, week 13
  validated child report of resilience; range: 12-60, higher scores reflect greater resilience
Brief Resilience Scale | week 0, week 13
  validated adult report of resilience; range 1-5, higher scores reflect greater resilience

CONTACTS AND LOCATIONS:
Overall Officials: Susana R Patton, PhD, Principal Investigator — Nemours Children's Health
Locations (2):
- United States (2):
  - Nemours Children's Health, Jacksonville, Florida
  - Children's Mercy Kansas City, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No